CLINICAL TRIAL: NCT03636438
Title: A Long-Term Follow-up Study to Evaluate Safety and Efficacy of Adeno-Associated Virus (AAV) Serotype 8 (AAV8)-Mediated Gene Transfer of Human Ornithine Transcarbamylase (OTC) in Adults With Late-Onset OTC Deficiency
Brief Title: Long Term Follow Up to Evaluate DTX301 in Adults With Late-Onset OTC Deficiency
Acronym: CAPtivate
Status: Active, not recruiting | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 301OTC02; 2018-000156-18 (EudraCT Number); 2022-501146-30-00 (EU CTIS Number)
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Ornithine Transcarbamylase (OTC) Deficiency
Keywords: gene therapy; OTC Deficiency; Urea Cycle Disorder
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease; Urea Cycle Disorders, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Determine the long-term safety of DTX301 following a single intravenous (IV) dose in adults with late-onset ornithine transcarbamylase (OTC) deficiency.

DETAILED DESCRIPTION:
Study 301OTC02 is a long-term follow-up study to evaluate the safety and efficacy of adeno-associated virus (AAV) serotype 8 (AAV8)-mediated gene transfer of human OTC in adults with late-onset OTC deficiency. Only subjects who complete Study 301OTC01 (NCT02991144) are eligible to participate in Study 301OTC02.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the Week 52 visit in Study 301OTC01.
2. Willing and able to provide written informed consent.
3. Willing, able, and committed to comply with scheduled study site visits, study procedures, and requirements.

Exclusion Criteria:

1. Planned or current participation in another interventional clinical study that may confound the efficacy or safety evaluation of DTX301 during the duration of this study.
2. Any clinically significant medical condition that, in the opinion of the investigator, would pose a risk to subject safety or would impede the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or older with OTC previously enrolled in Study 301OTC01
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events and Serious Adverse Events | Up to 416 weeks

SECONDARY OUTCOMES:
Change from Baseline Over Time in the Ureagenesis Rate | Baseline (average of Screening and Day 1) up to 416 weeks following DTX301 administration
  Sodium acetate is used as a tracer to measure the rate of ureagenesis
Change from Baseline Over Time in 24-Hour Area Under the Curve for Plasma Ammonia | Baseline (Day 0 of Study 301OTC01) up to 208 weeks following DTX301 administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceuticals Inc
Locations (9):
- United States (4):
  - The Children's Hospital Colorado, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Icahn School of Medicine, New York, New York
  - University Hospital Cleveland Medical Center/Case Western Reserve University, Cleveland, Ohio
- M.A.G.I.C. Clinic, Calgary, Alberta, Canada
- Hopital Femme Mere Enfant, Bron, Rhone, France
- Spain (2):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Coruna
  - Hospital Universitario de Cruces. Servicio de Pediatria, Barakaldo, Vizcaya
- Queen Elizabeth Hospital, Department of Endocrinology, Birmingham, United Kingdom

REFERENCES:
- See also: Ultragenyx Ornithine Transcarbamylase (OTC) Deficiency Research Study Opportunity — https://www.ultraclinicaltrials.com/OTC/
- See also: Ultragenyx Transparency Commitment — http://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/